CLINICAL TRIAL: NCT00852241
Title: Rejuvenation of the Lower Eyelid Using a Combination of Two Hyaluronic Acid Fillers - a Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF4
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Infraorbital Hollows
MeSH Terms: interventions — Hyaluronic Acid; Perlane

ARMS (1):
- Restalyne and Perlane (Experimental): One syringe of Perlane® (1.0cc) and one syringe of Restylane® (1.0cc) will be used total for both tear trough areas.
  Interventions: Drug: Restalyne; Drug: Perlane

INTERVENTIONS:
Drug: Restalyne — one syringe of Restylane® (1.0cc) will be used total for both tear trough areas.
  Other Names: Hyaluronan; Hyaluronate Sodium; Hyaluronic Acid
Drug: Perlane — One syringe of Perlane® (1.0cc) will be used total for both tear trough areas.
  Other Names: Hyaluronan; Hyaluronate Sodium; Hyaluronic Acid

SUMMARY:
The primary objective of this study is to determine the efficacy and longevity of the use of Restylane® and Perlane® in combination for the rejuvenation of the infraorbital hollows and to measure patient satisfaction with this treatment

DETAILED DESCRIPTION:
This study will examine the effectiveness of using Restylane® and Perlane® together in the treatment of the hollows in the under eye area. The combination of these treatments for use in the under eye area is considered investigational. An investigational therapy is a therapy that is not approved by the US Food and Drug Administration (FDA). Restylane® and Perlane® has been approved for treatment of moderate to severe facial wrinkles and folds, such as nasolabial folds by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* No significant medical illness
* Subjects with the willingness and ability to understand and provide informed consent

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or Lactation
* Subjects who have had previous surgical treatment of the lower eyelid area or previous use of filling agents in the under eye area
* Subjects with a known allergy to the components in Restylane® or Perlane®
* Subjects currently taking blood thinners or who have had chemotherapy or radiation within the last 6 months
* Subjects with liver/kidney disease or compromise or who are immunocompromised
* Subjects with a known susceptibility to keloid formation or hypertrophic scarring
* Subjects with an open, non-healing sore or infection near the site of injections
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Tung, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Restalyne and Perlane: One syringe of Perlane® (1.0cc) and one syringe of Restylane® (1.0cc) will be used total for both tear trough areas.
  Restalyne and Perlane: One syringe of Perlane® (1.0cc) and one syringe of Restylane® (1.0cc) will be used total for both tear trough areas.
Period: Overall Study
Arm/Group | Restalyne and Perlane
Started | 18
Completed | 0
Not Completed | 18
Not completed — Physician Decision | 18

BASELINE CHARACTERISTICS:
Population: The Principal Investigator left the institution and no data is available.
Arm/Group | Restalyne and Perlane
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants] — Population: PI left institution no data is available.
Sex/Gender, Customized [Count of Participants; unit: Participants] — female only. PI left institution, no data is available. Population: PI left institution, no data is available.

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Study is to Determine the Efficacy and Longevity of the Use of Restylane® and Perlane® in Combination for the Rejuvenation of the Infraorbital Hollows and to Measure Patient Satisfaction With This Treatment
Time Frame: 1 year
Population: The Principle Investigator left the institution and no data is available.
Arm/Group | Restalyne and Perlane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Restalyne and Perlane
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
PI left institution, no data is available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes